CLINICAL TRIAL: NCT02648789
Title: Validation of DNA Methylation Biomarkers for Oral Cancer Detection
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: iStat Biomedical CO., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-06-009AC
Record Dates: First submitted 2015-11-19; First posted 2016-01-07 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2017-05

CONDITIONS: Oral Cancer; Recurrence
Keywords: Primary oral cancer; DNA methylation; Recurrence oral cancer
MeSH Terms: conditions — Mouth Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — oral swab, non-cancerous matched tissue and tumor tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the correlation between DNA methylation and the treatment and recurrence of oral cancer.

DETAILED DESCRIPTION:
In this study, investigators plan to recruit 40~50 patients who had, or currently has oral cancer. The study procedures are as below:

* After the Informed Consent Form is signed, swab from the lesion site and normal site to obtain oral epithelial cells.
* Collect tissue from the tumor site and the non-cancerous matched site from the surgery or the tissue bank.
* Collect oral swab from the lesion site and the normal site when patients return to the clinic for a regular follow-up.

Specimens will be collected for DNA methylation testing, and the results will be compared with patient's clinical diagnosis. It is expected that the relationship between DNA methylation, oral cancer, and the recurrence of oral cancer will be found.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 75 years old
* Had or currently has cancer of the oral cavity
* Agree to sign the Informed Consent Form (ICF) and comply with follow-up procedures

Exclusion Criteria:

* Unwilling to sign the Informed Consent Form (ICF)
* Has an autoimmune disease of the oral cavity

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators plan to retrieve the tissue from the biobank in Taipei Veterans General Hospital or recruit oral cancer patients in this study over six months. The total patient number are 40-50. Specimen types include non-cancerous matched tissues, cancer tissues, and the oral swab. DNA methylation for several genes will be tested by using standardized reagents and instruments.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Association between the DNA methylation level and the stage of cancer | 1 year
  1. Compare the DNA methylation level and the stage of cancer before treatment.
  2. DNA methylation level as a monitor tool for recurrence/metastasis of oral cancer.
  3. qPCR will be used to determine the DNA methylation level.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chieh Yang, DDS., Ph.D., Principal Investigator — Department of Stomatology, Taipei Veterans General Hospital; Shou-Yen Kao, DDS., M.D.S., Principal Investigator — Department of Stomatology, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Wang SS, Smiraglia DJ, Wu YZ, Ghosh S, Rader JS, Cho KR, Bonfiglio TA, Nayar R, Plass C, Sherman ME. Identification of novel methylation markers in cervical cancer using restriction landmark genomic scanning. Cancer Res. 2008 Apr 1;68(7):2489-97. doi: 10.1158/0008-5472.CAN-07-3194. PMID 18381458
- [Background] Sova P, Feng Q, Geiss G, Wood T, Strauss R, Rudolf V, Lieber A, Kiviat N. Discovery of novel methylation biomarkers in cervical carcinoma by global demethylation and microarray analysis. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):114-23. doi: 10.1158/1055-9965.EPI-05-0323. PMID 16434596
- [Background] Lai HC, Lin YW, Chang CC, Wang HC, Chu TW, Yu MH, Chu TY. Hypermethylation of two consecutive tumor suppressor genes, BLU and RASSF1A, located at 3p21.3 in cervical neoplasias. Gynecol Oncol. 2007 Mar;104(3):629-35. doi: 10.1016/j.ygyno.2006.10.003. Epub 2006 Nov 13. PMID 17097722
- [Background] Towle R, Garnis C. Methylation-mediated molecular dysregulation in clinical oral malignancy. J Oncol. 2012;2012:170172. doi: 10.1155/2012/170172. Epub 2012 May 7. PMID 22645611
- [Background] Garcia MP, Garcia-Garcia A. Epigenome and DNA methylation in oral squamous cell carcinoma. Methods Mol Biol. 2012;863:207-19. doi: 10.1007/978-1-61779-612-8_12. PMID 22359295
- [Background] Nagata S, Hamada T, Yamada N, Yokoyama S, Kitamoto S, Kanmura Y, Nomura M, Kamikawa Y, Yonezawa S, Sugihara K. Aberrant DNA methylation of tumor-related genes in oral rinse: a noninvasive method for detection of oral squamous cell carcinoma. Cancer. 2012 Sep 1;118(17):4298-308. doi: 10.1002/cncr.27417. Epub 2012 Jan 17. PMID 22252571
- [Background] Fakhry C, Gillison ML. Clinical implications of human papillomavirus in head and neck cancers. J Clin Oncol. 2006 Jun 10;24(17):2606-11. doi: 10.1200/JCO.2006.06.1291. PMID 16763272
- [Background] Chaturvedi AK, Engels EA, Anderson WF, Gillison ML. Incidence trends for human papillomavirus-related and -unrelated oral squamous cell carcinomas in the United States. J Clin Oncol. 2008 Feb 1;26(4):612-9. doi: 10.1200/JCO.2007.14.1713. PMID 18235120
- [Background] Huang YK, Peng BY, Wu CY, Su CT, Wang HC, Lai HC. DNA methylation of PAX1 as a biomarker for oral squamous cell carcinoma. Clin Oral Investig. 2014 Apr;18(3):801-8. doi: 10.1007/s00784-013-1048-6. Epub 2013 Aug 2. PMID 23907469